CLINICAL TRIAL: NCT01279356
Title: Analysis of Volatile Organic Compounds in Exhaled Air as a Non-invasive Biomarker for Liver Diseases
Brief Title: Volatile Organic Compounds (VOCs) and Liver Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. dr. A. Masclee, Maastricht University Medical Center
Other Study IDs: MEC 10-3-088
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Liver Diseases
Keywords: Liver diseases; Volatile organic compounds; Inflammation; Oxidative stress; non-invasive tests
MeSH Terms: conditions — Liver Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following biospecimens will be collected: exhaled air and plasma/serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with liver diseases of various etiologies: * viral hepatitis
  * cholestatic liver diseases
  * auto-immune hepatitis
  * NAFLD
  * ALD
  * sarcoidosis of the liver

SUMMARY:
Liver diseases such as non-alcoholic fatty liver disease (NAFLD), alcoholic liver disease (ALD) and viral hepatitis have the potential to progress to cirrhosis and finally hepatocellular carcinoma (HCC). Early diagnosis and treatment of liver diseases is important since progression is likely and is associated with significant morbidity and mortality. However, in daily clinical practice no specific and non-invasive biomarkers are used for the diagnosis and follow-up of patients with liver diseases. It is known that patients with liver diseases produce compounds that can be excreted in breath as a consequence of metabolic processes, inflammation and/or oxidative stress. These are called volatile organic compounds (VOCs). Analysis of VOCs in exhaled air has been reported to provide valuable information in patients with chronic obstructive lung disease (COPD) and inflammatory bowel disease (IBD). Also, in patients with liver disease, exhaled VOCs have been detected.

The investigators hypothesize that analysis of VOCs in exhaled air of patients with liver diseases can be used for diagnosis and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of liver diseases based on laboratory, radiological and histological characteristics
* Age between 18 and 85 years

Exclusion Criteria:

* Inflammatory bowel disease
* Chronic obstructive lung disease, lung cancer, asthma
* Rheumatoid arthritis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with various liver diseases visiting the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To establish the validity of VOC analysis in exhaled air to discriminate between liver diseases and non-diseased controls | 12 months

SECONDARY OUTCOMES:
To compare the VOC profiles in exhaled air between various liver diseases | 12 months
To compare the VOC analysis before, during and after therapeutic interventions in various liver diseases | 12 months
To compare VOC profiles with systemic inflammatory and oxidative stress markers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Division of Gastroenterology/Hepatology, Maastricht, Limburg, Netherlands